CLINICAL TRIAL: NCT01029080
Title: Dynamic Cerebrovascular Autoregulation During Sepsis and Sepsis-associated Delirium
Brief Title: Cerebrovascular Autoregulation During Sepsis
Status: Completed | Type: Observational
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Patrick Schramm, Senior Physician, Johannes Gutenberg University Mainz
Other Study IDs: 837.435.08
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2013-04

CONDITIONS: Sepsis; Delirium
Keywords: Brain, blood flow; Measurement techniques, flow velocity waveform analysis; Monitoring, intensive care; Sepsis; transcranial doppler ultrasound (TCD); Cerebrovascular autoregulation; sepsis-associated delir
MeSH Terms: conditions — Sepsis; Delirium

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sepsis: All patients with sepsis defined by actually sepsis guidelines
  Interventions: Other: no interventions

INTERVENTIONS:
Other: no interventions — No interventions

SUMMARY:
The aim of the study is to correlate the dynamic cerebrovascular autoregulation by patients with sepsis with a sepsis-associated delirium.

ELIGIBILITY:
Inclusion Criteria:

* clinical symptoms of sepsis, severe sepsis and septic shock
* possibility for measurement of transcranial doppler ultrasound
* age over 18 years

Exclusion Criteria:

* preexisting cerebrovascular disease
* preexisting immunological disease
* traumatic brain injury
* intracranial infectious disease
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients at intensive care unit were screened to symptoms that definate sepsis
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-12; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Disturbed cerebrovascular autoregulation correlates with sepsis associated delir | 1 year
  The Index of autoregulation (Mx) was measured and correlated with the clinical incidence of a sepsis associated delir

SECONDARY OUTCOMES:
Correlation between inflammatory parameters and disturbed cerebrovascular autoregulation | 1 year
Correlation between inflammatory parameters and sepsis-associated delirium | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- University medical centre Mainz, Mainz, Germany

REFERENCES:
- [Result] Schramm P, Klein KU, Falkenberg L, Berres M, Closhen D, Werhahn KJ, David M, Werner C, Engelhard K. Impaired cerebrovascular autoregulation in patients with severe sepsis and sepsis-associated delirium. Crit Care. 2012 Oct 4;16(5):R181. doi: 10.1186/cc11665. PMID 23036135